CLINICAL TRIAL: NCT03049150
Title: The Use of Urinary MALDI-MS in Predicting Post-Operative Acute Kidney Injury in Patients After Fixation of Fractured Neck of Femur.
Brief Title: PREdicting RENAL Injury In Patient After Hip Fracture Surgery
Acronym: PRE-RENAL
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC16138
Record Dates: First submitted 2017-02-08; First posted 2017-02-09 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Acute Kidney Injury
Keywords: Urine; Mass Spectometry; Observational
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine whether MALDI, a type of Mass-Spectometry, can use protein pattern detection within urine to predict postoperative (after an operation) kidney damage in adults who have undergone emergency hip fracture surgery?

DETAILED DESCRIPTION:
The PRE-RENAL study is a prognostic accuracy study testing the ability of the MALDI-MS assay to predict incident acute kidney injury after fractured neck of femur surgery. The study aims to validate the findings of a urinary peptide panel previously developed and validated on a cohort of septic patients.

Kidney injury following surgery or as a part of severe illness is an important complication, because it can delay and reduce the chances of recovery. A reliable early test for kidney injury would be useful so that treatments to prevent or minimise it can be started as early as possible. This study, based with a group of medical researchers working with chemists, will analyse clinical urine specimens from patients undergoing major orthopaedic (bone) surgery. We will explore whether patterns of proteins in the urine could be used as an early warning that kidney injury is present before existing tests demonstrate it.

ELIGIBILITY:
Inclusion Criteria:

* Fractured Neck of Femur
* Age >50
* Informed consent

Exclusion Criteria:

* Refusal of Consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 50 years old who have suffered fractured neck of the femur
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | Within 7 days
  Defined by KDIGO Criteria

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No